CLINICAL TRIAL: NCT05883631
Title: Prospective, Single Arm, Multi-center, Clinical Evaluation of the Ablacath™ Mapping Catheter and Ablamap® System Utilizing Electrographic Flow (EGF) Mapping to Resolve Extra-pulmonary Vein Sources of Atrial Fibrillation and Guide Ablation Therapy.
Brief Title: RESOLVE-AF: Clinical Evaluation of the Ablacath™ Mapping Catheter and Ablamap® System Utilizing Electrographic Flow (EGF) Mapping to Resolve Extra-PV Sources of Atrial Fibrillation and Guide Ablation Therapy.
Acronym: RESOLVE-AF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cortex (Industry)
Collaborators: Ablacon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP006
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation, Persistent; Atrial Fibrillation Paroxysmal; Arrhythmia; Arrhythmias, Cardiac; Atrial Flutter; Atrial Fibrillation, Paroxysmal or Persistent; Atrial Arrhythmia; Atrial Tachycardia
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- De Novo Arm: Electrographic Flow (EGF) mapping (Experimental): Subjects with persistent or long-standing persistent atrial fibrillation (AF), coming in for a De Novo pulmonary vein isolation procedure.
  Interventions: Device: Electrographic Flow (EGF) mapping (no ablation)
- Redo Arm: Electrographic Flow (EGF) mapping and guided ablation of EGF-identified sources (Experimental): Subjects with paroxysmal, persistent or long-standing persistent atrial fibrillation (AF) coming in for a redo AF procedure.
  Interventions: Device: Electrographic Flow (EGF) mapping and ablation of EGF-identified sources of Atrial Fibrillation

INTERVENTIONS:
Device: Electrographic Flow (EGF) mapping and ablation of EGF-identified sources of Atrial Fibrillation — In addition to standard touch-up of pulmonary vein isolation, subjects receive targeted source ablation guided by Electrographic Flow™ (EGF) mapping. EGF mapping enables the full spatiotemporal reconstruction of organized atrial electrical wavefront propagation to identify active sources or origins of excitation that may trigger atrial fibrillation (AF).
  EGF-identified sources with activity above the threshold (≥ 25%) are considered significant and targeted with radiofrequency ablation. The procedure concludes when all EGF-identified sources are eliminated, defined as reducing source activity below the threshold.
  Other Names: OptiMap™ System
  Arms: Redo Arm: Electrographic Flow (EGF) mapping and guided ablation of EGF-identified sources
Device: Electrographic Flow (EGF) mapping (no ablation) — In addition to standard pulmonary vein isolation (PVI), subjects receive Electrographic Flow™ (EGF) mapping. PVI may be performed using any commercially available platform/catheter.
  EGF mapping enables the full spatiotemporal reconstruction of organized atrial electrical wavefront propagation to identify active sources or origins of excitation that may trigger atrial fibrillation (AF). EGF-identified sources with activity above the threshold (≥ 25%) are marked as relevant; however, no EGF-guided ablations are performed during this index procedure. If subjects have AF recurrence after the 90-day blanking period, they may undergo a recurrence procedure and EGF-guided ablation.
  Other Names: OptiMap™ System
  Arms: De Novo Arm: Electrographic Flow (EGF) mapping

SUMMARY:
Demonstrate the safety and effectiveness of the Ablacath™ Mapping Catheter and Ablamap® System in patients with all types of atrial fibrillation (AF) including paroxysmal or persistent or long-standing persistent, undergoing and De Novo or Redo procedures.

Phenotype patients and demonstrate the prognostication power of Electrographic Flow (EGF®) maps among all subjects using 12-month follow-up outcomes following EGF-guided mapping and ablation.

DETAILED DESCRIPTION:
Subjects with all types of AF who are candidates for catheter ablation of their AF. The study will enroll up to 400 subjects in 25 centers globally.

ELIGIBILITY:
Inclusion Criteria:

1. Suitable candidate for intra-cardiac mapping and ablation of atrial arrhythmias including atrial fibrillation, atrial flutter and/or atrial tachycardia
2. Above eighteen (18) years of age or of legal age to give informed consent specific to state and national law
3. Left atrial (LA) diameter ≤ 5.5 cm or LA volume index ≤ 50 mL/m2 (use whichever measure is available or if both available, use the lesser of the two to qualify)

Exclusion Criteria:

1. De Novo paroxysmal AF
2. AF from a reversible cause (e.g., surgery, hyperthyroidism, sarcoidosis, or pericarditis, etc.)
3. Cardiac surgery or intervention within the past 90 days (e.g. percutaneous coronary intervention, ablation for ventricular arrhythmias, left atrial appendage occlusion devices, atrial septal defect closure devices, transcatheter aortic valve replacement)
4. Presence of transvenous pacing or defibrillator leads or an atrial leadless pacemaker
5. Myocardial infarction within the past 90 days
6. Severe valvular disease or prosthetic valve(s)
7. Contraindication to therapeutic anticoagulation
8. Decompensated heart failure or New York Heart Association (NYHA) Functional Class IV
9. Positive pregnancy test
10. Any other contraindication to an intracardiac mapping and ablation of atrial arrhythmias
11. Enrollment in another investigational study evaluating another device, biologic or drug

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with 12-month freedom from AF recurrence (with or without AADs) | From 90 days to 12 months after index procedure
  This measure represents the number of subjects with freedom from documented episodes of atrial fibrillation (AF) recurrence lasting longer than 30 seconds from the 90-day post-procedure blanking period through 12 months of follow-up (with or without AADs).
Number of participants with freedom from a composite of serious adverse events (SAEs) occurring within 7 days from the index procedure | From index procedure to 7 days after index procedure
  Evaluated by assessing combined rate of SAE composite as adjudicated by a CEC for relatedness to device or procedure
Demonstrate the predictive value of electrographic flow (EGF) phenotyping for ablation outcome | 12 months

SECONDARY OUTCOMES:
Number of participants with freedom from a composite of SAE occurring within 30 days from post-index ablation procedure | From index procedure to 30 days after index procedure
  Evaluated by assessing combined rate of SAE composite as adjudicated by a CEC for relatedness to device or procedure
Overall reduction in burden of AF for subset of patients with implantable loop recorder | From 90 days to 12 months after index procedure
  Evaluation of patient's freedom from AF based on recordings of implantable loop recorders
Overall procedure time, fluoro time, total EGF-guided mapping time, total EGF-guided ablation time | Index or Repeat Procedure
  Evaluation of index or recurrence procedure data

CONTACTS AND LOCATIONS:
Overall Officials: Kent Nilsson, MD, Principal Investigator — Piedmont Athens Regional; Lucas Boersma, Prof. MD., Principal Investigator — St. Antonius Hospital
Locations (24):
- United States (15):
  - University of Alabama, Birmingham, Alabama
  - Grandview Medical Center, Birmingham, Alabama
  - Banner Health, Phoenix, Arizona
  - Sutter Health Sequoia Heart and Vascular Institute, Redwood City, California
  - Pacific Heart Institute, Santa Monica, California
  - Colorado Heart, Golden, Colorado
  - Florida Heart Rhythm Specialists, Fort Lauderdale, Florida
  - Ascension Medical Group, Jacksonville, Florida
  - Piedmont Health, Athens, Georgia
  - Beaumont Health, Royal Oak, Michigan
  - Mount Sinai Hospital, New York, New York
  - Ohio State University, Columbus, Ohio
  - University of Virginia, Charlottesville, Virginia
  - Inova Health, Falls Church, Virginia
  - Evergreen Health Research/Overlake Medical Center, Bellevue, Washington
- Belgium (3):
  - OLV Hospital Aalst, Aalst
  - ZNA Middelheim, Antwerp
  - ZOL, Genk
- Czechia (3):
  - Neuron Medical, Brno
  - IKEM (Institute for Clinical and Experimental Medicine), Prague
  - Na Homolce Hospital, Prague
- Netherlands (3):
  - Amsterdam UMC (location AMC), Amsterdam, North Holland
  - St. Antonius Hospital, Nieuwegein, Utrecht
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: No